CLINICAL TRIAL: NCT02484053
Title: Implementation of Rapid Infusion Rituximab in a Pilot Group of Adolescents With Hematologic, Oncologic, and Rheumatologic Disorders
Brief Title: Rapid Infusion Rituximab, Hematologic, Oncologic, and Rheumatologic Disorders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jenny Despotovic, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-35628 Rituximab
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Hematologic Disorders; Oncologic Disorders; Rheumatologic Disorders
Keywords: adult and pediatric cancers; blood disorders; lymphoma; graft-versus-host-disease; diseases of the immune system
MeSH Terms: conditions — Hematologic Diseases; Lymphoma; Graft vs Host Disease | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rheumatologic disease (Experimental): Rituximab is administered over 120 minutes, 12.5% of the dose will be given over the first 30 minutes and the remaining 87.5% of the dose will be given over 90 minutes.
  Interventions: Drug: Rituximab
- Cancer or blood disorder (Experimental): Rituximab is administered over 90 minutes, 20% of the dose will be given over the first 30 minutes and the remaining 80% of the dose will be given over 60 minutes.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Giving rituximab as a rapid infusion over a period of 90 or 120 minutes.

SUMMARY:
Rituximab is frequently used in adult and pediatric cancers, blood disorders, lymphoma (a cancerous growth made up of lymphoid tissue), graft-versus-host-disease (complication that can occur after a stem cell or bone marrow transplant), diseases of the immune system (the cells and substances that protect the body from infection) and rheumatologic conditions. Rituximab works by decreasing or temporarily eliminating a specific type of white blood cell, the B-lymphocyte. Overall, rituximab is generally well tolerated. The likelihood of an infusion-related reaction, or symptoms such as fever, chills, hives, low blood pressure or swelling, is very low, but highest during a patient's first infusion of rituximab and decreases with each additional dose. Adults commonly receive rituximab at a faster rate if they have done well with the first infusion, this study will help determine if the same approach is well tolerated in children.

In this study, the investigators are testing a new method of administering rituximab which may reduce the time it takes to receive the medication. The initial ordered amount of rituximab will not change from the current standard of care (meaning what is usually done by doctors, and would likely be done if you were not on this study). The period of time over which rituximab is given is what is being studied.

DETAILED DESCRIPTION:
The standard of care in patients receiving rituximab is to give the dose slowly and gradually increase the rate of rituximab until the full dose is given, which may take several hours. This is done in order to prevent a side effect of rituximab called an infusion reaction. Infusion reactions are similar to allergic reactions and may cause symptoms such as low blood pressure, wheezing, chest tightness, fever, itching, bad cough, blue skin color, seizures, or swelling of the face, lips, tongue, or throat.

In this study, the investigators are testing the method of giving rituximab over a shorter period of time. Administering rituximab at this faster rate is done commonly and safely in the adult population with very few side effects.

The drug rituximab will be given as an infusion in the outpatient clinic. Infusion means the drug is given using a needle or tubing inserted into a vein (also called an IV) over a period of time.

If patients have a cancer or blood disorder, they will receive rituximab administration over 90 minutes, 20% of the dose will be given over the first 30 minutes and the remaining 80% of the dose will be given over 60 minutes. This is the standard method of infusing doses of rituximab in adults who have a cancer or blood disorder, and have done well with a first dose of rituximab at the standard infusion rate.

If patients have a rheumatologic disease, they will receive rituximab administration over 120 minutes, 12.5% of the dose will be given over the first 30 minutes and the remaining 87.5% of the dose will be given over 90 minutes. This is the standard method of infusing doses of rituximab in adults who have a rheumatologic disorder, and have done well with a first dose of rituximab at the standard infusion rate.

During this time, the investigator will also assess to see if patients have any side effects from receiving the faster infusion and for 15 minutes following the end of the infusion. Patients will also be followed up by phone or in clinic one week after the rapid infusion of rituximab to see if they have any side effects.

Before patients receive rituximab, they will receive acetaminophen and diphenhydramine. These medications are given to help prevent an infusion reaction from occurring. These medications are always given no matter how quickly rituximab is given.

If an infusion reaction occurs, the rituximab infusion will stop and patients will receive medications to help reverse the reaction. Once the reaction has gone away, the patient's doctor will determine if and how they will receive the rest of their rituximab dose.

Patients will receive one rapid infusion of rituximab as part of their participation in this study. If patients did not have an infusion-related reaction they are eligible to receive subsequent infusions off protocol at the discretion of the provider.

Patients will be asked to allow us to view and collect information from their medical records prior to their infusion to ensure eligibility and obtain baseline data, as needed on the day of their infusion and through the next clinical follow up to monitor for side effects from the infusion. Data collected from the medical records includes but is not limited to, demographic information (age, race/ethnicity, weight, diagnoses, and indication for rituximab).

ELIGIBILITY:
Inclusion Criteria:

* Previously received and tolerated at least one rituximab infusion via standard infusion administration. *No modifications or adjustment to the infusion, or treatment with any anaphylaxis reaction medications required
* No history of Grades 3 or 4 infusion reaction to rituximab based on the NIH Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
* Prescribed rituximab with the following indications and doses for administration in the outpatient setting:

  * Hematologic or oncologic indication: 100 mg/m^2 or 375 mg/m^2
  * Rheumatologic indication: 375-750 mg/m^2 (total dose not to exceed 1000 mg)

Exclusion Criteria:

* Any patient not meeting the inclusion criteria.
* Any patient who does not consent to the pilot protocol.
* Any patient on a clinical trial where the infusion rate of rituximab is prescribed by the clinical trial.
* Any patient who required rescue or symptomatic treatment with steroids, antihistamines, or epinephrine during prior rituximab infusions.
* Any patient who has received a bone marrow transplant.

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety of rapid infusion rituximab in a pilot group of adolescent patients for hematologic, oncologic, and rheumatologic disorders. | 6 weeks
  To be measured by the administration of rapid infusion rituximab without requiring modifications to therapy as a result of adverse reactions

SECONDARY OUTCOMES:
To determine the incidence of infusion-related reactions with the administration of rapid infusion rituximab | 6 weeks
  To be measured as the number of patients who experience a grade 3 or higher infusion-related reaction

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Despotovic, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States